CLINICAL TRIAL: NCT03105986
Title: A Phase 1, Randomized, Open-label, Crossover Study to Evaluate the Effect of the Organic Anion Transporter Inhibitor Probenecid on the Pharmacokinetics of JNJ-64041575 in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Effect of the Organic Anion Transporter Inhibitor Probenecid on the Pharmacokinetics of JNJ-64041575 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108300; 64041575RSV1002 (Other: Janssen-Cilag International NV); 2016-003923-49 (EudraCT Number)
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Participants will receive Treatment A (1000 milligram (mg) oral dose of JNJ-64041575 on Day 1) in Period 1, followed by Treatment B (1000 mg oral dose of JNJ-64041575 on Day 22 along with probenecid 500 mg on Day 21 to Day 28) in Period 2. A washout Period of 21 days will be maintained between each Period.
  Interventions: Drug: JNJ-64041575; Drug: Probenecid
- Treatment sequence BA (Experimental): Participants will receive Treatment B (1000 mg oral dose of JNJ-64041575 on Day 1 along with probenecid 500 mg on Day -1 to Day 7) in Period 1, followed by Treatment A (1000 mg oral dose of JNJ-64041575 on Day 22) in Period 2. A washout Period of 21 days will be maintained between each Period.
  Interventions: Drug: JNJ-64041575; Drug: Probenecid

INTERVENTIONS:
Drug: JNJ-64041575 — Two 500-mg tablets administered as a single oral dose under fasted conditions on Day 1 or Day 22.
Drug: Probenecid — One 500-mg tablet administered as a single oral dose with a total of 30 doses (2 doses on Day -1/21 starting in the evening followed by 4 doses per day on the rest of the days).

SUMMARY:
The purpose of this study is to evaluate the effect of multiple-dose administration of probenecid on the pharmacokinetics of JNJ-63549109 and JNJ-64167896 after a single dose of JNJ-64041575 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI; weight in [Kilogram] kg divided by the square of height in meters) between 18.0 and 30.0 kilogram per meter square (kg/m^2, extremes included, and a body weight not less than 50.0 kg, inclusive, at screening
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in the protocol
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, extremes included, and no higher than 90 mmHg diastolic. If blood pressure is out of range, 1 repeated assessment is permitted after an additional 5 minutes of rest
* Participants must have normal values for alanine transaminase (ALT) and aspartate aminotransferase (AST) (less than or equal to [<=]1.0 × upper limit of normal [ULN])
* A female participant, except if postmenopausal, must have a negative serum beta human chorionic gonadotropin (Beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 and Day 21

Exclusion Criteria:

* Participant has a history of current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease (example: glucose-6-phosphate-dehydrogenase deficiency), coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness, that in the investigator's and/or sponsor's medical monitor opinion should exclude the participant or that could interfere with the interpretation of the study results
* Participants with 1 or more of the following laboratory abnormalities at screening as defined by the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table: [1] Serum creatinine grade 1 or greater (>1.0 × [Upper Limit of Normal] ULN) [2] Hemoglobin grade 1 or greater (<=10.5 grams per deciliter [g/dL]) [3] Platelet count grade 1 or greater (<=99,999/ cubic millimeter [mm^3]) [4] Reticulocyte count (absolute) below the lower limit of laboratory normal range [5] Absolute neutrophil count grade 1 or greater (<=1,500/mm^3) [6] Total bilirubin grade 1 or greater (>1.0 × ULN) [7] Any other toxicity grade 2 or above, except for grade 2 elevations of low density lipoprotein cholesterol and/or cholesterol
* Participants with a history of uric acid kidney stones, conditions associated with elevated urinary uric acid excretion, participants with peptic ulcer disease or a history of peptic ulcer disease, or other contra-indications for the use of probenecid
* Participants has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  Cmax is the maximum observed plasma concentration.
Area Under Plasma Concentration Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of JNJ-63549109 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  Area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-63549109 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-64167896 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  Cmax is the maximum observed plasma concentration.
Area Under Plasma Concentration Time Curve From Time Zero to the Last Quantifiable (AUC [0-last]) of JNJ-64167896 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  Area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64167896 (Metabolite of JNJ-64041575) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | From Signing of Informed Consent Form (ICF) to End of Study (Approximately up to 88 days)
  An adverse event is any untoward medical event that occurs in a subject administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany